CLINICAL TRIAL: NCT02138812
Title: An Open-label Phase I Dose-escalation Study to Characterize the Safety, Tolerability, Pharmacokinetics, and Maximum Tolerated Dose of Oral BAY1161909 in Combination With Weekly Intravenous Paclitaxel Given in an Intermittent Dosing Schedule in Subjects With Advanced Malignancies
Brief Title: Phase I Dose Escalation of Oral BAY1161909 in Combination With Intravenous Paclitaxel
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: As another Mps1 inhibitor was being developed in parallel, the strategic decision was to move forward with the development of the follow up compound only.
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 16804
Record Dates: First submitted 2014-05-08; First posted 2014-05-15 (Estimated); Last update posted 2018-10-12 (Actual); Status verified 2018-10

CONDITIONS: Medical Oncology
Keywords: Phase 1; Solid tumors; Breast cancer; Paclitaxel; Mps-1 inhibitor; Taxanes
MeSH Terms: conditions — Breast Neoplasms | interventions — Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- BAY1161909 + Paclitaxel (Experimental): Participants received oral doses of BAY1161909 starting from 0.75 mg twice daily, from C1D1 onwards in a 2 days on/5 days off dosing schedule as single agent treatment in Cycle 1 (14 days), and from C2D8 onwards in a 2 days on/5 days off dosing schedule in combination with weekly intravenous paclitaxel on D1, D8, and D15 of the 28-day cycles. For single-dose Pharmacokinetic (PK) cohort: in Cycle 1, participants received a single oral dose of 6 mg BAY1161909 on C1D1 with no BAY1161909 dosing for the remainder of Cycle 1.
  Interventions: Drug: BAY1161909; Drug: Paclitaxel

INTERVENTIONS:
Drug: BAY1161909 — Given orally, with a starting dose of 0.75 mg twice daily from C1D1 onwards in a 2 days on/5 days off dosing schedule as single agent treatment in Cycle 1 (14 days), and from C2D8 onwards in a 2 days on/5 days off dosing schedule in 28-day cycles. For single-dose PK cohort: a single oral dose on C1D1
Drug: Paclitaxel — 75 mg/m^2 (initial dose escalation) or 90 mg/m^2 (second dose escalation), weekly intravenously (IV) infusion on D1, D8, and D15 of the 28-day cycles from C2D1

SUMMARY:
Determine the safety, tolerability, maximum tolerated dose (MTD), and recommended Phase II dose (RP2D) of BAY1161909 in combination with paclitaxel in subjects with advanced malignancies.

DETAILED DESCRIPTION:
BAY1161909 is a potent and highly selective inhibitor of monopolar spindle 1 (Mps1) kinase activity. Human Mps1 is a serine threonine kinase which functions as a core component of the spindle assembly checkpoint (SAC), a key surveillance mechanism that monitors the attachment of spindle microtubules to the kinetochores of the chromosomes during pro-metaphase and halts the transitions to anaphase until all chromosomes are bi-oriented, fully attached, and correctly tensed at the metaphase plate. Mps1 is expressed in the mitosis phase of the cell cycle in proliferating cells. Overexpression of Mps1 has been observed in several cancer cell lines and tumor types including lung and breast cancers.

Established anti-mitotic drugs such as vinca alkaloids, taxanes, or epothilones activate the SAC either by destabilizing or stabilizing spindle microtubules resulting in mitotic arrest. Prolonged arrest in mitosis forces a cell either into a mitotic exit without cytokinesis or into a mitotic catastrophe leading to cell death. In contrast, Mps1 inhibitors inactivate the SAC and accelerate progression of cells through mitosis eventually resulting in severe chromosomal missegregation, mitotic catastrophe, and cell death. Consequently, Mps1 inhibition leads to failure of cells to arrest in mitosis in response to anti-mitotic drugs. Thus, the combination of microtubule-interfering agents and Mps1 inhibition strongly increases chromosomal segregation errors and cell death and therefore, constitutes an efficient strategy for selectively eliminating tumor cells.

This study will attempt to answer the following questions:

* What are the side effects of BAY1161909 when given at different dose levels and schedules with paclitaxel?
* What dose level and schedule of BAY1161909 should be tested in future clinical research studies?
* How much BAY1161909 and paclitaxel is in the blood at specific times after administration?
* Does the treatment with BAY1161909 with paclitaxel show any effect on the tumor growth?
* Are there specific biomarkers that might be able to explain why some patients respond to treatment and others do not.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects aged =/> 18 years
* Subjects with advanced, histologically or cytologically confirmed advanced malignancies (solid tumors), refractory to any standard therapy, have no standard therapy available, or subjects actively refused any standard treatment and / or if, in the judgment of the investigator, experimental treatment is clinically and ethically acceptable.
* For the expansion cohort: women with histologically or cytologically confirmed triple negative breast cancer (TNBC)
* Subjects must have evaluable or measurable disease according to Response Evaluation Criteria In Solid Tumors (RECIST) 1.1
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 1
* Life expectancy of at least 12 weeks
* Adequate bone marrow, liver, and renal functions

Exclusion Criteria:

* Known hypersensitivity to the study drugs or excipients of the preparations or any agent given in association with this study
* Evidence of peripheral neuropathy of Grade > 2
* History of cardiac disease: congestive heart failure New York Heart Association (NYHA) class > II, unstable angina (anginal symptoms at rest), new-onset angina (within the past 3 months before study entry), myocardial infarction within the past 3 months before study entry, or cardiac arrhythmias requiring anti-arrhythmic therapy (beta blockers, calcium channel blockers, and digoxin are permitted)
* Prior treatment with more than 3 lines of cytostatic therapies for metastatic disease unless specifically agreed between investigator and sponsor. Subjects with a history of any prior Grade =/> 3 toxicity associated with taxane treatment will be excluded.
* Uncontrolled hypertension defined as systolic blood pressure >150 mmHg or diastolic blood pressure >90 mmHg, despite optimal medical management
* Moderate or severe hepatic impairment, i.e. Child-Pugh class B or C
* History of human immunodeficiency virus (HIV) infection.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 69 (Actual)
Dates: Start 2014-05-09 (Actual); Primary Completion 2017-04-28 (Actual); Study Completion 2017-10-02 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose (MTD) | Up to 2 years
  MTD is defined as the highest dose of oral BAY1161909 (administered in combination with or without IV paclitaxel) that can be given such that not more than 30% of the subjects experience a dose-limiting toxicity (DLT) during Cycles 1 and 2. The safety profile of oral BAY1161909 will first be determined in combination with 75 mg/m^2 IV paclitaxel [MTD (75)]. Starting in >Cohort 7 (12 mg 2 times daily [BID] BAY1161909) the MTD of oral BAY1161909 will then be refined for the combination with 90 mg/m^2 IV paclitaxel [MTD (90)].
Number of subjects with adverse events and serious adverse events as a measure of safety and tolerability. | Up to 2 years
Plasma concentration of Paclitaxel characterized by Cmax | C2D1 (without oral BAY1161909): pre-dose and 0.5,1,2,3,4,6,8,12,24 (C2D2) & 48hrs (C2D3) after the start of IV infusion on C2D1. C2D8 (with oral BAY1161909): pre-dose and 0.5,1,2,3,4,6, 8,12,24 (C2D9) & 48hrs (C2D10) after the start of infusion on C2D8.
Plasma concentration of BAY1161909 characterized by Cmax | C1D1: pre-dose & 0.5,1,2,3,4,6,8,12 hrs after the MD on C1D1 [12-hour sample to be collected before administration of the ED]. C1D2: pre-dose & 0.5,1,2,3,4,6,8,12, 24 (C1D3), 48 (C1D4), 72 (C1D5) & 144 hrs (C1D8 pre-dose) after the MD on C1D2.
  C1D1 (single-dose PK without IV paclitaxel), C1D2 (multiple-dose PK without IV paclitaxel; no ED on C1D2, MD=Morning Dose, ED= Evening Dose
Plasma concentration of BAY1161909 characterized by Cmax | C2D8 (single-dose PK with IV paclitaxel): pre-dose and 0.5, 1, 2, 3, 4, 6, 8, 12 hours after the morning dose on C2D8 [12-hour sample to be collected before administration of the evening dose].
Plasma concentration of BAY1161909 characterized by Cmax | C1D1 (single-dose PK cohort only): pre-dose and 0.5, 1, 2, 3, 4, 6, 8, 12, 24 (C1D2), 48 (C1D3), 72 (C1D4), 96 (C1D5), 168 (C1D8), 240 (C1D11) and 336 hours (before C2D1 IV paclitaxel administration) after the morning dose on C1D1.
Plasma concentration of BAY1161909 characterized by Cmax | C1D-7 (relative bioavailability assessment subjects): pre-dose and 0.5, 1, 2, 3, 4, 6, 8, 12, 24 (C1D-6), and 72 (C1D-4) hours after the single dose on C1D-7.

OTHER OUTCOMES:
Tumor response evaluation following RECIST 1.1 criteria | Up to 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (6):
- United States (6):
  - Santa Monica, California
  - New Haven, Connecticut
  - Boston, Massachusetts
  - Detroit, Michigan
  - Nashville, Tennessee
  - San Antonio, Texas